CLINICAL TRIAL: NCT05495347
Title: Big Data Analysis of OSA Patients on Positive Airway Pressure (PAP) Treatment: Real-life Monitoring: TeleVAL Study
Brief Title: Big Data Analysis of OSA Patients on Positive Airway Pressure (PAP) Treatment: Real-life Monitoring
Acronym: TeleVAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Other Study IDs: TeleVAL
Record Dates: First submitted 2022-08-05; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Obstructive Sleep Apnea; Positive Airway Pressure
Keywords: telemonitoring; big data
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Registry of patients
  Interventions: Other: patients diagnosed with OSA

INTERVENTIONS:
Other: patients diagnosed with OSA — All patients diagnosed with OSA since March 2020 with an indication for treatment with PAP have been telemonitored permanently since the start of therapy and continue to be telemonitored at the present time. Data are sent remotely daily to the telemonitoring platform.

SUMMARY:
The present study aims to determine to what extent remote monitoring of PAP related to patients' clinical parameters is able to provide relevant data on predictors of compliance, subgroups of patients who may benefit from this technological tool, variations in AHI over time, occurrence of central events at the start of therapy and, in short, to shed new light on this disease and its treatment, all within the application of continuous positive pressure therapy in the real world.

Among the intended objectives is the identification of phenotypes involved in the use and efficacy of PAP therapy: development of a predictive model, as well as the evaluation of the impact of long-term telemonitoring of patients with Obstructive Sleep Apnea (OSA).

The study initially arose from the need to diagnose, treat and follow up patients with suspected OSA in compliance with the social distancing rules imposed by the COVID-19 pandemic.

It is an ambispective cohort study, with retrospective data collection from the start date of the pandemic (March 2020) to December 2021, and prospective data collection from the approval of the protocol to December 2022.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with OSA since March 2020 with indication for treatment with PAP have been telemonitored on an ongoing basis since initiation of therapy continuing to be telemonitored at the current time.

Exclusion Criteria:

* Undiagnosed OSA patients

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Obstructive Sleep Apnea (OSA)
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterize the phenotypes involved | pandemic start date March 2020 until December 2022.
  Determine the emergent CSA appearance in relation to PAP treatment.

SECONDARY OUTCOMES:
Establish the percentage of patients who at the first connection to the TM achieved the optimal therapeutic pressure | pandemic start date March 2020 until December 2022.
  According to Built in software (BIS) of the equipment
Establish the Profile of patients who at the first connection to the TM achieved the optimal therapeutic pressure | pandemic start date March 2020 until December 2022.
  According to Built in software (BIS) of the equipment
Variations in AHI during the first year of follow-up and their relationship with patient characteristics. | pandemic start date March 2020 until December 2022.
Time to achieve the optimal therapeutic pressure described after the first connection | pandemic start date March 2020 until December 2022.
  Number of modifications required and their relationship with patient subgroups.
Evaluation of the impact of long-term telemonitoring of patients with OSA | pandemic start date March 2020 until December 2022.
  Number of acesses and interventions made to the telemonitoring platform/year and time invested

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Marques de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No